CLINICAL TRIAL: NCT01402583
Title: Menopause is a Critical Factor in Determining Failure of Antiviral Therapy in Women With Chronic Hepatitis C - An Epidemiological Study
Brief Title: Menopause is a Critical Factor in Determining Failure of Antiviral Therapy in Women With Chronic Hepatitis C
Acronym: MEN_EPID
Status: Completed | Type: Observational
Sponsor: Prof. Facchinetti Fabio (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Prof. Facchinetti Fabio, Prs admin, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: RSO-321
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Gender; Menopause; Sustained viral response; Cytokines
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Coitus | interventions — Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEG IFN/Ribavirin: Subjects with Hepatitis C undergoing PEG IFN/Ribavirin treatment
  Interventions: Drug: PEG IFN/Ribavirin

INTERVENTIONS:
Drug: PEG IFN/Ribavirin — PEG IFN/Ribavirin
  Other Names: Pegylated IFN 2a Pegasys; Pegylated IFN 2b PegIntron; Copegus; Rebetol

SUMMARY:
Menopause represents a critical period in a woman's life as the hormonal changes and the failing ovarian function not only determine relevant modifications in the reproductive function but also in many other conditions and organs that apparently are scarcely linked with hormones. The PI's centre has among its main goals the treatment of chronic liver disease; in the last years, a increasing interest in gender-related issues has grown.

Goal of this study is to verify the impact of menopause on response to antiviral therapy for CHC and in determining more severe fibrosis in comparison with age-matched men. To achieve this goal a database of all the PEG IFN/Ribavirin patients treated in the GI Unit of the University of Modena and Reggio Emilia in the last 7 years will be set up. Demographic, clinical and biochemical data as well data regarding the reproductive history, time, type, length of estrogen deprivation and of hormone-replacement therapy will be collected.

DETAILED DESCRIPTION:
The study is designed retrospective epidemiological cohort study. Overall, a group of 442 women (168 still in fertile age; 274 menopausal) with HCV-positive CAH who underwent PEG IFN treatment in the last 5 years will be evaluated. For comparison, a group of 548 HCV-positive males with CAH will be evaluated. Liver biopsies before undergoing standard antiviral therapy will be scored for fibrosis, inflammation and steatosis. In women the presence, type and timing of menopause, associated hormonal/metabolic features and serum interleukin-6 (IL-6) and hepatic tumor necrosis factor-α (TNF-α) levels will be evaluated.

The primary endpoint will be evaluation of SVR in females (in fertile and menopausal age) and in males.

ELIGIBILITY:
Inclusion Criteria:

* All women treated for HCV chronic hepatitis, at the Unit Gastroenterology, University of Modena and Reggio Emilia, in the last 7 years.
* Control group is a cohort matched for age (ratio 1:1) selected from a group of 558 men with chronic HCV treated in the same period

Exclusion Criteria:

* No exclusion criteria aret pre-defined as the study includes all patients who were treated for chronic HCV hepatitis; exclusion was made upstream of the constitution of this cohort.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of 442 women (168 still in fertile age; 274 menopausal) with HCV-positive CAH who underwent PEG IFN treatment in the last 5 years will be evaluated. For comparison, a group of 548 HCV-positive males with CAH will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ERICA VILLA, Prof, Principal Investigator — University of Modena & Reggio Emilia
Locations (1):
- Gastroenterology Unit, Modena, Italy